CLINICAL TRIAL: NCT03989908
Title: Insulinemic and Glycemic Evaluation of Microfluidic Food Grade Gel in Food Applications.
Brief Title: Effects of Microfluidic Noodle on Blood Glucose Levels of Healthy Volunteers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Health System (Unknown)
Responsible Party: Principal Investigator, Mei Hui Liu, Principal Investigator, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/01062
Record Dates: First submitted 2019-06-17; First posted 2019-06-18 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: microfludic
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study is a within-subject cross-over trial design to assess the glycemic response of microfluidic noodle consumption by human subjects as compared to mee sua (control noodle).
Who Masked: Participant
Masking Description: Participants are blinded to the noodles served.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Co-flow alginate/SPI food gel (Experimental): Direction of flow in alginate and SPI are in the same direction in the production of the microfluidic noodle.
  Interventions: Other: Microfludic noodle
- Counter-flow alginate/SPI food gel (Experimental): Direction of flow in alginate and SPI are in the opposite direction in the production of the microfluidic noodle.
  Interventions: Other: Microfludic noodle
- Mee Sua (Placebo Comparator): Mee Sua is used as a control to compare the outcome due to its similarity in textural properties
  Interventions: Other: Control noodle

INTERVENTIONS:
Other: Microfludic noodle — In this intervention arm, subjects will be served with noodles made using microfludic technology.
  Arms: Co-flow alginate/SPI food gel; Counter-flow alginate/SPI food gel
Other: Control noodle — In this intervention arm, subjects will be served with normal noodle.
  Arms: Mee Sua

SUMMARY:
In this study, microfluidics was applied in the creation of low-GI food gel made from non-traditional ingredients like alginate and soy protein isolate. This method is previously tested to produce lower glycaemic response than normal noodle and pasta.

DETAILED DESCRIPTION:
Research has confirmed that a food's glycemic effect cannot be accurately predicted from the type and amount of carbohydrates it contains, as the rate at which the carbohydrates is digested and released into the bloodstream is influenced by many factors such as the food's physical form, its fat, protein and fibre content, and the chemical structure of its carbohydrates. For these reasons, it is possible to produce food from the same group with different effects on blood glucose. Consumption of low GI food has shown to improve glycemic control, lipid profile and reduce systemic inflammation. However, there are few dietary intervention studies attempting to change the GI of food by changing the staple carbohydrates. In this study, microfluidics was applied in the creation of low-GI food gel made from non-traditional ingredients like alginate and soy protein isolate. This method is previously tested to produce lower glycaemic response than normal noodle and pasta. With noodles being one of the staples to many Singaporeans, food gels formed using functional ingredients derived from food sources offer a lower GI alternative to the conventional noodle and pasta without affecting the people dietary preference.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Age between 21-65 years old
* Overtly healthy males or females, as determined by medical history, physical examination and laboratory results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Males and females with stable medical problems that, in the investigator's opinion, will not significantly alter the performance of the biomarker panel, will not place the subject at increased risk by participating in the study, and will not interfere with interpretation of the data.
* Not on any regular medications (western / traditional medicine). Nutritional supplements with established chemical composition that can be ascertained and clearly recorded is acceptable.
* Have venous access sufficient to allow for blood sampling as per the protocol
* Reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Body mass index range of 18-25kg/m2 for male and 18-23kg/m2 for female.

Exclusion Criteria:

* History or presence of current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, malignancy or neurological disorders capable of significantly altering the performance of the biomarker panel; or of interfering with the interpretation of data
* Known or ongoing psychiatric disorders within 3 years
* Regularly use known drugs of abuse within 3 years
* Women who are pregnant or lactating
* Have donated blood of more than 500 mL within 4 weeks of study enrolment
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females):

  * 1 unit = 12 oz or 360 mL of beer;
  * 5 oz or 150 mL of wine;
  * 1.5 oz or 45 mL of distilled spirits
* Uncontrolled hypertension (blood pressure [BP] >160/100mmHg
* Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
* Treatment with any investigational drug, or biological agent within one (1) month of screening or plans to enter into an investigational drug/ biological agent study during the duration of this study
* Known allergy to insulin
* History of bleeding diathesis or coagulopathy
* Any of the following laboratory values at screening:

Fasting glucose >=126mg/dL(>=7mmol/L) or 2 hour post-prandial glucose >=200mg/dL (>=11.1mmol/L)

* Clinically significant (as determined by investigator) abnormalities on laboratory examination that will increase risk to the patient or interfere with data integrity
* Have any other conditions, which, in the opinion of the Investigator would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the study
* Significant change in weight (+/- 5%) during the past month
* Allergy to test food

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-13 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in glucose response | 2 hour
  A meal tolerance test will be done to collect blood samples for glucose analysis at 0 min, 15 min, 30 min, 45 min, 60 min , 90 min and 120 min.The change in glucose response will be measured by comparing incremental area under the curve (iAUC) after ingestion of Microfluidic noodle meal and control Mee sua meal.
Change in insulin response | 2 hour
  A meal tolerance test will be done to collect blood samples for glucose analysis at 0 min, 15 min, 30 min, 45 min, 60 min , 90 min and 120 min.The change in insulin response will be measured by comparing incremental area under the curve (iAUC) after ingestion of Microfluidic noodle meal and control Mee sua meal.

SECONDARY OUTCOMES:
Change in ghrelin level | 2 hour
  A meal tolerance test will be done to collect blood samples for glucose analysis at 0 min, 30 min, 60 min , 90 min and 120 min.The change in ghrelin level will be measured by comparing AUC after ingestion of Microfluidic meal and control Mee sua meal.
Change in glucagon-like peptide 1 (GLP-1) level | 2 hour
  A meal tolerance test will be done to collect blood samples for glucose analysis at 0 min, 30 min, 60 min , 90 min and 120 min.The change in GLP-1 level will be measured by comparing AUC after ingestion of Microfluidic meal and control Mee sua meal.
Change in satiety rating | 2 hour
  A visual analogue scale (VAS) will be presented to the participants at 0, min, 30 min, 60 min , 90 min and 120 min, to indicate how they feel in response to 4 given statements by marking an "X" on a 100-mm line.
  At time T=12 min, palatability of the treatment was assessed by five characteristics, from bad (0 mm) to good (100 mm). These characteristics were visual appeal, smell, taste, texture, and overall pleasantness of the meal given. Scores were determined by measuring the distance (in mm) from the let starting point of the line to the intersection of the "X". Subjects did not discuss their ratings.The primary outcome was area under the curve (AUC) for responses on the VAS calculated using the trapezoidal rule.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Hui Liu, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
The plan for individual participant data will be discussed with collaborator to decide whether to be shared.